CLINICAL TRIAL: NCT00002283
Title: Randomized Prospective Study of Dapsone Versus Trimethoprim-Sulfamethoxazole in the Treatment of First Episode Pneumocystis Carinii Pneumonia in AIDS Patients
Brief Title: A Comparison of Dapsone and Trimethoprim-Sulfamethoxazole in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobus Pharmaceutical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 007A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Dapsone; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Trimethoprim; Sulfamethoxazole; Dapsone

INTERVENTIONS:
Drug: Trimethoprim
Drug: Sulfamethoxazole
Drug: Dapsone

SUMMARY:
Evaluate the effectiveness rate of dapsone plus trimethoprim as a therapy for the first episode of Pneumocystis carinii pneumonia (PCP) in AIDS patients. Compare the rates and severity of adverse effects using dapsone versus trimethoprim - sulfamethoxazole (TMP / PurposeX). Establish relative toxicities with regard to suitability for outpatient treatment.

ELIGIBILITY:
Exclusion Criteria

Concurrent Medication:

Excluded:

* Requirement for other medications found to be effective in the treatment of Pneumocystis carinii pneumonia (PCP) (i.e., DFMO, pyrimethamine, and sulfadiazine).

Patients with the following are excluded:

* History of allergic reaction to dapsone.
* Requirement for other medications found to be effective in the treatment of Pneumocystis carinii pneumonia (PCP) (i.e., DFMO, pyrimethamine, and sulfadiazine).
* Patients subsequently found to be glucose-6-phosphate dehydrogenase (G6PD) positive will be withdrawn from the study and treated with another regimen.

Prior Medication:

Excluded:

* Requirement for other medications found to be effective in the treatment of Pneumocystis carinii pneumonia (PCP) (i.e., DFMO, pyrimethamine, and sulfadiazine).

Patients who are glucose-6-phosphate dehydrogenase (G6PD) positive will be withdrawn from the study and treated with another regimen.

Hospitalized patients with first episode of Pneumocystis carinii pneumonia (PCP) documented by GIEMSA or methenamine stain.

* Patients must:
* Be willing and able to give informed consent.
* Be expected to survive 1 week without therapy.
* Have less than 48 hours of treatment for Pneumocystis carinii pneumonia (PCP) for this episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobus Pharmaceutical Co, Princeton, New Jersey, United States